CLINICAL TRIAL: NCT02352649
Title: 1-2 Phase of Safety and Efficacy of Patient Intraneural Injections of VEGF165 Plasmid Gene Therapy on Regeneration After Total Severance or Disruption of the Entire Nerve Fiber
Brief Title: Safety and Efficacy Study of Neovasculgen (Pl-VEGF165) Gene Therapy in Patients With Peripheral Nerve Injury
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Artgen Biotech (Other)
Collaborators: Kazan Federal University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Neurotmesis
Record Dates: First submitted 2015-01-24; First posted 2015-02-02 (Estimated); Last update posted 2015-02-02 (Estimated); Status verified 2015-01

CONDITIONS: Peripheral Nerve Injury
Keywords: Peripheral nerve injury; Neurotmesis; Gene therapy; Plasmid; Nerve regeneration therapy
MeSH Terms: conditions — Peripheral Nerve Injuries; Trauma, Nervous System

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Neovasculgen 1 (Experimental): Gene therapy drug Neovasculgen will be administered by several intraneural injections after surgical nerve reconstruction before wound closing. A dose is 0,6 mg will be dissolved in 1 ml of aqueous vehicle (water for injection) prior to injection.
  Interventions: Drug: Neovasculgen
- Neovasculgen 2 (Experimental): Gene therapy drug Neovasculgen will be administered by several intraneural injections after surgical nerve reconstruction before wound closing. A dose is 1,2 mg will be dissolved in 1 ml of aqueous vehicle (water for injection) prior to injection.
  Interventions: Drug: Neovasculgen
- water for injections (Placebo Comparator): Instead of the gene therapy drug, 1 ml of aqueous vehicle (water for injections) will be administered by several intraneural injections.

INTERVENTIONS:
Drug: Neovasculgen
  Arms: Neovasculgen 1; Neovasculgen 2

SUMMARY:
The purpose of this study is to determine safety and efficacy of pl-vegf165 ("Neovasculgen") for regeneration of peripheral nerve. Pl-vegf165 ("Neovasculgen") is the permitted in Russian Federation angiogenic medication that induce growth of new vessels and included in a complex therapy for patients with peripheral arterial diseases in Russia. It has also been shown to enhance nerve regeneration and muscle reinnervation in animals but these properties have not previously been studied in patients. Moreover, currently there is no method in clinical use to speed the rate of recovery after nerve injury. The objective of this study is to explore the ability of pl-vegf165 to benefit the treatment of patients with peripheral nerve injury. The investigators hypothesize that treatment with intraneural injections with pl-vegf165 after peripheral nerve reconstruction will accelerate nerve regeneration, reduce the period of denervation and improve muscle reinnervation and recovery in patients with peripheral nerve injury.

DETAILED DESCRIPTION:
All patients enrolled into the study will receive standard surgery procedures indicated in accordance with medical care standards for the certain disease. Patients after nerve injury classified as neurotmesis will receive surgical repair of injured nerves what will be added by intraneural injections of pl-vegf165. Safety and efficacy of gene therapy will be assessed by physical examination, comprehensive laboratory tests over next 18 month after surgical nerve reconstruction.

ELIGIBILITY:
Inclusion Criteria:

* Patients with confirmed transection injury between shoulder and wrist
* Isolated injury of ulnar or median nerve (not mixed injury of several nerves)
* Nerve injuries which are amenable to direct end-to-end repair
* Length of the gap between of stumps of transected nerve no longer than 3,5 centimeters
* Early delayed (secondary) repair performed between 2 to 6 weeks after nerve injury

Exclusion Criteria:

* Length of the gap between of stumps of transected nerve more than 3,5 centimeters
* Simultaneous injury of several peripheral nerves
* Localization of nerve injury beyond of forearm
* Presence of neurological deficit preceding to nerve injury
* Systemic disease of connective tissue
* Myopathy
* Large surgical procedures planned for next one and a half year
* Presence of oncological diseases
* Pregnancy and breastfeeding
* Alcohol and drug addiction
* Patient ability to adhere strictly to the rules of the current clinical trial protocol

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2015-04; Primary Completion 2016-03 (Estimated); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
Disabilities of the Arm, Shoulder and Hand (DASH) Measure | 540 days
  The Disabilities of the Arm, Shoulder and Hand (DASH) Outcome Measure is a 30-item, self-report questionnaire designed to measure physical function and symptoms in patients with any or several musculoskeletal disorders of the upper limb. The questionnaire was designed to help describe the disability experienced by people with upper-limb disorders and also to monitor changes in symptoms and function over time. Testing has shown that the DASH performs well in both these roles.
Adverse events | 540 days

SECONDARY OUTCOMES:
Medical Research Council (MRC) Scale for Muscle Strength | 90 days;180 days; 270 days; 360 days; 450 days; 540 days
  In this scale, muscle strength is graded on a scale from 0 to 5 depending on ability to make whole fall active range of motion and presence of muscle resistance
The Short Form (36) Health Survey | 90 days;180 days; 270 days; 360 days; 450 days; 540 days
  The SF-36 consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability. The higher the score the less disability i.e., a score of zero is equivalent to maximum disability and a score of 100 is equivalent to no disability.
Nerve conduction velocity | 180 days; 360 days; 540 days
  For electrodiagnostic assessment, nerve conduction velocity (NCV) was tested as motor and sensory. The results categorized according to the Yale sensory scale and the severity of sensation and function of the nerves was scored as follows: 0, no sensation; 1, decreased or abnormal sensation; 2, normal sensation.
Electromyography | 180 days; 360 days; 540 days
  For an EMG, a needle electrode was inserted through the skin into the muscle which injured nerve supplied. The presence, size and shape of the waveform registered and the ability of the muscle to respond when the nerves were stimulated. Also these results scored as follows: 0, no activity; 1, few or single movement; 2, partial activity; 3, full activity.